CLINICAL TRIAL: NCT02970435
Title: Evaluating the Impact of Video Discharge Instructions for Mohs Surgery Post-Operative Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1616
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Linear Closure; Surgery
Keywords: surgery; video discharge instructions
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Discharge Instructions (Experimental): These videos contain the same instructions that a patient receives via the standard-of-care verbal and written discharge instructions. These instructions will be delivered by the same nursing and medical staff that also regularly provides verbal and written discharge instructions to patients. There will be no difference in the content between the standard-of-care verbal and written instructions and the video discharge instructions. Patients in this group will receive telecommunication reminders on how to access discharge videos.
  Interventions: Behavioral: Video Discharge Instructions; Behavioral: Telecommunication Reminders; Behavioral: Standard of Care
- Verbal and Written Discharge Instructions (Active Comparator): Nursing and medical staff will provide verbal and written discharge instructions as is standard of care post surgery
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Video Discharge Instructions — The video discharge instructions, will be provided to the patient at the time of surgical procedure.
  Arms: Video Discharge Instructions
Behavioral: Telecommunication Reminders — Telecommunication reminders including text messages, email, or phone calls to remind participants how to access the video discharge instruction up to three times before follow-up
  Arms: Video Discharge Instructions
Behavioral: Standard of Care — Standard of Care: verbal and written discharge instructions for patients after surgery

SUMMARY:
The purpose of this research is to look at how educational videos provided by doctors might affect patients knowledge, satisfaction, confidence, and anxiety with post-operative Mohs surgery care. Patients will be randomized to either: 1) a group that receives educational videos in addition to standard-of-care written and verbal instructions or 2) a group that receives only standard-of-care written and verbal instructions.

DETAILED DESCRIPTION:
The Primary Objective of this study is to determine if video discharge instructions, when added to standard of care written and verbal instructions, lead to a decrease in unnecessary phone calls from patients in a Mohs dermatology clinic.

The Secondary Objectives of this study are to determine if video discharge instructions, when added to standard of care written and verbal instructions, help to improve patients' satisfaction with education materials provided by the clinic, improve patients' knowledge of post-operative management, improve patients' confidence in taking care of their suture site post-operatively, and reduce post-operative anxiety about their suture site.

This study will be a randomized controlled trial in which the impact of video discharge instructions on patient calls, anxiety, and confidence will be evaluated. Patients will be randomized using a permuted block model generated through SAS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a linear closure on the face at UH Mohs clinic
* Fluent English speakers

Exclusion Criteria:

● Non-fluent English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Ratio of patients in the intervention group who call the clinic compared to percentage of patients in the control group who call the clinic | Up to 8 weeks after discharge
  Researchers will record when each participant calls the clinic. The number of people who call in the intervention group will be compared to the number of people who call in the control group. This will give an efficacy measure of the video discharge instructions

SECONDARY OUTCOMES:
Difference in knowledge of discharge instructions in intervention group versus control group | Up to 8 weeks after discharge
  Answers to survey questions investigating knowledge of discharge instruction will be compared between the control and intervention groups.
Difference in confidence in intervention group versus control group | Up to 8 weeks after discharge
  A survey investigating confidence about Mohs surgery post-operative care will be used in this study. This survey will be quantified using the Likert scale.
Difference in satisfaction in intervention group versus control group | Up to 8 weeks after discharge
  A survey investigating patient satisfaction about Mohs surgery post-operative care will be used in this study. This survey will be quantified using the Likert scale.
Difference in self reported anxiety levels in intervention group versus control group | Up to 8 weeks after discharge
  A survey investigating anxiety about Mohs surgery post-operative care will be used in this study. This survey will be quantified using the Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Bordeaux, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals at Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States